CLINICAL TRIAL: NCT07040917
Title: A Study to Evaluate the Safety and Efficacy of CAR-T Cells in Subjects With Autoimmune Diseases
Brief Title: A Study of CAR-T Cells in Subjects With Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhu, Clinical Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AID01
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Diseases
Keywords: autoimmune diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment (Experimental)
  Interventions: Drug: CAR-T cell

INTERVENTIONS:
Drug: CAR-T cell — CAR-T cell

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CAR-T cell therapy in Subjects with autoimmune diseases.

DETAILED DESCRIPTION:
This is a single center, one-arm, open label study aiming to evaluate the safety and efficacy of CAR-T cells therapy in subjects with autoimmune diseases.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, between 18 and 65 years old;
2. Diagnosed with Autoimmune Diseases, such as Systemic Lupus Erythematosus, Systemic Sclerosis, Idiopahic Inflammatory Myopathies, Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis, Sjögren's Syndrome, Antiphospholipid Syndrome, Immune Thrombocytopenia, Pemphigus；
3. Good organ functions;
4. Subjects must understand and personally, voluntarily sign and date an informed consent.

Key Exclusion Criteria:

1. Had or has active malignancy;
2. Patients who have previously received CD19-targeted drugs, or CAR-T therapy, or any other gene therapy products;
3. Combined with other autoimmune disease that needs systemic treatment or therapy;
4. Pregnant or lactating women;
5. Has other factors that deemed not suitable by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 0~28 day after treatment
Frequency of adverse events, serious adverse events | within 24 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China